CLINICAL TRIAL: NCT03339778
Title: An Investigator Driven Observational Study to Determine the Benefit of Octagam 5% for Treatment of Patients Diagnosed With Primary Immunodeficiency Disorders (PID) on Intravenous Immunoglobulin (IVIG) Therapy That Experience Adverse Events (AEs) on Any 10% IVIG Preparation
Brief Title: The Benefit of 5% IVIG for Patients With Primary Immunodeficiency Disorders Who Experience Adverse Events on 10% IVIG Preparations
Status: Completed | Type: Observational
Sponsor: IMMUNOe Research Centers (Industry)
Responsible Party: Sponsor
Other Study IDs: IIS201401-PID
Record Dates: First submitted 2015-03-31; First posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Primary Immunodeficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patients with primary immunodeficiency disorders (PID) on intravenous immunoglobulin (IVIG) treatment may experience adverse events (AEs). Patients who experience AEs on any 10% IVIG solution will be changed to octagam 5% for six infusions to evaluate the potential benefit for reduction of AEs on a lower concentration IVIG product.

DETAILED DESCRIPTION:
Patients with PID require life long immunoglobulin (Ig) replacement therapy with IVIG being the most common form. As more 10% IVIG products are FDA approved, the older and well characterized 5% IVIG products are becoming less used. Currently, the standard of care for patients who experience AEs on IVIG is to move to a subcutaneous (SCIG) delivery and product. This study will evaluate the AEs on a 10% product and octagam 5%. The study will enroll 15 patients after an AE on any 10% product who will then be infused with octagam 5% for six infusions. AEs will be documented and compared to the 10% product along with changes in biomarkers. The study data may document another therapeutic option for patients who experience AEs - SCIG and octagam 5%.

ELIGIBILITY:
Inclusion Criteria:

* Participants, or legal guardians with assent by underage children, will sign informed consent/assent and are willing to comply with all aspects of the study
* Diagnosis of CVID according IUIS Expert Committee
* Participants on a 10% product who experience AEs
* Ages between 10 and 75 years of age
* Participants on 10% IVIG therapy every 21±3 days or 28±3 days between 300 - 800 mg/Kg body weight

Exclusion Criteria:

* Acute infection requiring antibiotic therapy within 7 days prior to visit 1
* Presence of any condition that is likely to interfere with the evaluation of the study medication or satisfactory conduct of the trial
* History of anaphylactic or severe systemic reactions to human immunoglobulin
* IgA deficient patients with antibodies against IgA and a history of hypersensitivity
* Females who are pregnant or lactating

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosis of PID - specifically common variable immunodeficiency (CVID)
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2015-06 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
The change in the number of AEs post-infusion between any 10% IVIG product and octagam 5% | AEs will be documented at screening and up to 72 hours post-infusion for six infusions up to 24 weeks

SECONDARY OUTCOMES:
The change in levels of inflammatory biomarkers associated with AEs between any 10% IVIG and octagam 5% | Levels will be documented at screening and up to 72 hours post-infusion for six infusions up to 24 weeks
Safety Evaluations (complete blood count [CBC]) | Screening and prior to each infusion (six infusions total) up to 24 weeks
  CBC
Safety evaluations (Complete Metabolic profile[CMP]) | Screening and prior to each infusion (six infusions total) up to 24 weeks
  CMP
Safety evaluations (IgG trough level) | Screening and prior to last infusion up to 24 weeks
  IgG trough level

CONTACTS AND LOCATIONS:
Overall Officials: Isaac Melamed, MD, Principal Investigator — IMMUNOe Research Centers

REFERENCES:
- [Background] Geha RS, Notarangelo LD, Casanova JL, Chapel H, Conley ME, Fischer A, Hammarstrom L, Nonoyama S, Ochs HD, Puck JM, Roifman C, Seger R, Wedgwood J; International Union of Immunological Societies Primary Immunodeficiency Diseases Classification Committee. Primary immunodeficiency diseases: an update from the International Union of Immunological Societies Primary Immunodeficiency Diseases Classification Committee. J Allergy Clin Immunol. 2007 Oct;120(4):776-94. doi: 10.1016/j.jaci.2007.08.053. PMID 17952897
- [Background] Deane S, Selmi C, Naguwa SM, Teuber SS, Gershwin ME. Common variable immunodeficiency: etiological and treatment issues. Int Arch Allergy Immunol. 2009;150(4):311-24. doi: 10.1159/000226232. Epub 2009 Jul 1. PMID 19571563
- [Background] Kaveri SV, Maddur MS, Hegde P, Lacroix-Desmazes S, Bayry J. Intravenous immunoglobulins in immunodeficiencies: more than mere replacement therapy. Clin Exp Immunol. 2011 Jun;164 Suppl 2(Suppl 2):2-5. doi: 10.1111/j.1365-2249.2011.04387.x. PMID 21466545
- [Background] Maarschalk-Ellerbroek LJ, Hoepelman IM, Ellerbroek PM. Immunoglobulin treatment in primary antibody deficiency. Int J Antimicrob Agents. 2011 May;37(5):396-404. doi: 10.1016/j.ijantimicag.2010.11.027. Epub 2011 Jan 26. PMID 21276714